CLINICAL TRIAL: NCT06327893
Title: Patients Treated by the Danish Emergency Medical Services Following Non-drowning Water Rescues From 2016 to 2023: A Danish Registry-based Study From 2016 to 2023
Brief Title: Patients Treated by the Danish Emergency Medical Services Following Non-drowning Water Rescues From 2016 to 2023
Acronym: RESCUE
Status: Recruiting | Type: Observational
Sponsor: Prehospital Center, Region Zealand (Other)
Responsible Party: Principal Investigator, Niklas Breindahl, Principel Investigator, Prehospital Center, Region Zealand
Other Study IDs: AQUATIC_RESCUE
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2024-03

CONDITIONS: Drowning; Drowning, Near; Submersion; Submersion - Accidental; Submersion or Drowning Due to Being Washed Overboard; Submersion or Drowning Due to Being Thrown Overboard; Submersion or Drowning Due to Ship Sinking, Water Skier Injured; Submersion or Drowning Due to Boat Submerging, Swimmer Injured; Submersion or Drowning Due to Boat Overturning, Swimmer Injured; Submersion or Drowning Due to Boat Submerging, Water Skier Injured; Submersion or Drowning Due to Fall From Gangplank, Swimmer Injured; Submersion or Drowning Due to Ship Sinking, Docker or Stevedore Injured; Submersion or Drowning Due to Fall Overboard, Docker or Stevedore Injured
Keywords: Water rescue; Aquatic rescue; Danish Prehospital Drowning Data; Danish Drowning Formula; Emergency Medical Service (EMS); Cohort; Registry; Utstein; Epidemiology
MeSH Terms: conditions — Drowning; Near Drowning | interventions — Immersion; Fluid Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Aquatic rescue: Patients treated by the Danish EMS following an aquatic rescue performed by lay or professional rescuers are identified from the Danish PEMR using the Danish Drowning Formula (DDF) and extensive manual validation.
  Interventions: Other: Submersion or immersion in liquid

INTERVENTIONS:
Other: Submersion or immersion in liquid — The patient must have been submersed or immersed in liquid.

SUMMARY:
Since 2015, all Danish prehospital EMS have used the nationwide Prehospital Electronic Medical Record (PEMR). In 2023, the investigators developed the Danish Drowning Formula (DDF), a text-search algorithm designed to search the unstructured text fields in the electronic medical records with comprehensive search criteria to identify all potential water-related incidents. This protocol describes the first study to analyse the prehospital data from a nationwide Danish cohort of patients treated by the EMS from 2016 to 2023 following non-drowning aquatic rescues.

DETAILED DESCRIPTION:
Purpose The purpose of this study is to establish recommendations towards specific educational, preventative, or rescue strategies to reduce the number of aquatic rescues in Denmark (e.g., campaigns targeting high-risk groups, or fencing, allocating rescue equipment, or establishing lifeguard stations in high-risk areas). This may not only enhance prevention of aquatic rescues but also decrease the mortality and the total number of drowning incidents in Denmark.

Objectives The primary objective is to estimate the yearly incidence of patients treated by the Danish EMS following a non-drowning aquatic rescue from 2016 to 2023 and calculate the aquatic rescue to drowning ratio. The secondary objectives are to characterise the rescues (e.g., lay rescuer or professional rescuer, use of equipment) and to report the spatial distribution.

Study design This study is a nationwide registry-based study with data from the Danish nationwide PEMR from 2016 to 2023.

Methods Since 2015, all Danish prehospital EMS have used the nationwide Prehospital Electronic Medical Record (PEMR). In 2023, the investigators developed the Danish Drowning Formula (DDF), a text-search algorithm designed to search the unstructured text fields in the electronic medical records with comprehensive search criteria to identify all potential water-related incidents. This study will be the first to analyse the prehospital data from a nationwide Danish cohort of patients treated by the EMS from 2016 to 2023 following non-drowning aquatic rescues.

ELIGIBILITY:
Inclusion Criteria:

* All the patients registered in the Danish Prehospital Electronic Medical Record from 2016-2023 will be screened by the Danish Drowning Formula and the medical records containing one or more trigger words will be extracted for manual validation.
* All records where the patient was immersed or submersed in liquid but did not experience mild, moderate, or severe respiratory impairment following the drowning process will be included.

Exclusion Criteria:

* All records where the patient was immersed or submersed in liquid and did experience mild, moderate, or severe respiratory impairment following the drowning process).
* All records where the patient was not immersed or submersed in liquid.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated by the Danish EMS following an aquatic rescue are identified from the Danish Prehospital Electronic Medical Record using the Danish Drowning Formula and extensive manual validation.
  We used the WHO definition of drowning supported by the "Clarification and Categorisation of Non-fatal Drowning" statement to differentiate between drowning and non-drowning aquatic rescues.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
The annual incidence. | From 2016 to 2023.
  The incidence will be reported as the annual number of cases.
The annual incidence rate. | From 2016 to 2023.
  The incidence rate will be reported as the annual number of cases per 100,000 person-years.

SECONDARY OUTCOMES:
The spatial distribution of aquatic rescues on a map of Denmark. | From 2016-2023.
  Each incident will be presented with a single entry based on the geographical coordinates of the incident.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Collatz Christensen, Ass. Prof., Study Director — Prehospital Center, Region Zealand
Locations (1):
- Prehospital Center, Næstved, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No
The datasets used and analysed during the current study are available from the corresponding author upon reasonable request.

REFERENCES:
- [Background] Breindahl N, Wolthers SA, Jensen TW, Holgersen MG, Blomberg SNF, Steinmetz J, Christensen HC; Danish Cardiac Arrest Group. Danish Drowning Formula for identification of out-of-hospital cardiac arrest from drowning. Am J Emerg Med. 2023 Nov;73:55-62. doi: 10.1016/j.ajem.2023.08.024. Epub 2023 Aug 15. PMID 37619443